CLINICAL TRIAL: NCT05032560
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics After Single and Multiple Doses of ABX464 Capsules in Healthy Japanese Volunteers.
Brief Title: Safety and Pharmacokinetics Study in Healthy Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-921
Record Dates: First submitted 2021-08-30; First posted 2021-09-02 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Part A: single-ascending-dose Part B: escalating multiple-dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 25 mg single dose (Experimental): Subject will receive a single oral dose of ABX464 25 mg or its matching placebo
  Interventions: Drug: ABX464; Drug: Placebo
- 50 mg single dose (Experimental): Subject will receive a single oral dose of ABX464 50 mg or its matching placebo
  Interventions: Drug: ABX464; Drug: Placebo
- 25 mg multiple dose (Experimental): Subject will receive a daily oral dose of ABX464 25 mg or its matching placebo for 28 days
  Interventions: Drug: ABX464; Drug: Placebo
- 50 mg mulptiple dose (Experimental): Subject will receive a daily oral dose of ABX464 50 mg or its matching placebo for 28 days
  Interventions: Drug: ABX464; Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — Drug: ABX464 ABX464 is a new anti-inflammatory drug
Drug: Placebo — Drug: Matching Placebo placebo matching with ABX464

SUMMARY:
The study consists of Part A, a randomized double-blind, single-ascending-dose study, and Part B, a randomized, double-blind, semi-sequential, escalating multiple-dose study, in healthy Japanese volunteers.

DETAILED DESCRIPTION:
Part A includes the following two dose regimen groups:

* 25 mg dose regimen group: ABX464 25 mg or placebo
* 50 mg dose regimen group: ABX464 50 mg or placebo In each dose regimen group, 12 subjects will be randomly assigned, according to a 3:1 ratio, to receive either ABX464 (9 subjects) or its matching placebo (3 subjects).

Part B includes the following two dose regimen groups:

* 25 mg dose regimen group: ABX464 25 mg or placebo for 28 days
* 50 mg dose regimen group: ABX464 50 mg or placebo for 28 days

In each dose regimen group, 12 subjects will be randomly assigned, according to a 3:1 ratio, to receive either ABX464 (9 subjects) or its matching placebo (3 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Male Japanese volunteers.
2. 20 to 45 years old.
3. Considered by the Investigator, as healthy based on history, physical examination, and complete laboratory evaluation (laboratory parameters should be within normal ranges of the study center's laboratory or considered not clinically significant by the Investigator).
4. Vital signs (supine blood pressure, resting pulse rate, body temperature) should be within normal ranges and no deviation from standard 12-lead electrocardiogram (ECG) should be observed at screening.

   Body mass index (BMI) should be between 18 (inclusive) and 27 kg/m² (inclusive).
5. Non-smokers at enrolment.
6. Subjects must understand, sign and date the written voluntary Informed Consent Form at the visit prior to any protocol-specific procedures.
7. Able and willing to comply with study visits and procedures as per protocol.
8. Males receiving the study treatment and their partners must agree to use a highly effective contraceptive method during the study and for 6 months after the last dose of study drug. Highly effective methods of contraception include true abstinence, intrauterine device (IUD) or hormonal contraception aiming at inhibition of ovulation, intrauterine hormone releasing system, bilateral tubal ligation, and vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the subject. In each case of delayed menstrual period (over 1 month between menstruations) in a female partner of a male subject, confirmation of absence of pregnancy of the partner is required. Male subjects must not be planning pregnancy, should use a condom and must not donate sperm during the study and for 6 months after the last dose of study drug.

Exclusion Criteria:

1. Acute disease state (e.g., nausea, vomiting, diarrhea, or fever within a week) or chronic infectious disease (positive results for hepatitis B surface antigen [HBsAg], hepatitis C virus antibody, human immunodeficiency virus antigen/antibody, tuberculosis determined by QuantiFERON-TB Gold Plus test). Subjects who have positive hepatitis B core antibody [HBcAb] can be enrolled but must have an undetectable hepatitis B virus [HBV] viral load (HBV DNA test).
2. Positive results for SARS-CoV-2 antigen determined by polymerase chain reaction method.
3. History of recent grade 3 or 4 opportunistic infection or underlying conditions that may predispose them to grade 3 or grade 4 infection.
4. History of cardiovascular, pulmonary, gastrointestinal, hepatic, pancreatic, renal, metabolic, hematological, neurological, psychiatric, or systemic disease that could jeopardize the safety of the subject or the validity of the study results.
5. Illicit drug or alcohol abuse, or dependence within a year.
6. Blood donation within 3 months prior to screening.
7. Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer.
8. Use of any immunosuppressive drugs (except topical steroids) within 3 months prior to first dose.
9. Any history of hypersensitivity to drugs.
10. Any condition, which in the opinion of the Investigator, could compromise the subject's safety or adherence to the study protocol

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and SAEs | 6 weeks
  number of incidences of all adverse events (AEs) (causally related and non-related) and SAEs, will be described further categorized by severity
incidence of treatment-emergent serious adverse events | 6 weeks
  number of incidences of treatment-emergent serious adverse events will be described
incidence of treatment-emergent adverse events of special interest (AESIs). | 6 weeks
  number of incidences of treatment-emergent adverse events of special interest (AESIs) will be described.
incidence of clinically significant laboratory abnormalities | 6 weeks
  number of incidences of clinically significant laboratory abnormalities will be described

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 42 days
  Cmax of ABX464 will be derived from the plasma concentrations
Area under the plasma concentration versus time curve (AUC) | 42 days
  AUC of ABX464 will be derived from the plasma concentrations
Time to reach the maximum plasma concentration (tmax) | 42 days
  Tmax of ABX464 will be derived from the plasma concentrations
miR124 level | 42 days
  concentration of miR124 expression will be measured in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No